CLINICAL TRIAL: NCT03907904
Title: Continuous, Non-invasive Monitoring of Intraoperative Cerebral Perfusion and Oxidative Metabolism (CPOM): a Knowledge Translation Study.
Brief Title: Continuous, Non-invasive Monitoring of Intraoperative Cerebral Perfusion and Oxidative Metabolism (CPOM)
Status: Completed | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: 113650
Record Dates: First submitted 2019-03-05; First posted 2019-04-09 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2020-10

CONDITIONS: Brain Hypoxia Ischemia
Keywords: Intraoperative/methods* Oximetry/methods* Oxygen/metabolism; brain/metabolism; brain chemistry; cerebrovascular circulation; humans; monitoring, intraoperative/methods; oximetry/methods; oxygen/metabolism
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CPOM Optical Neuromonitor — Prior to induction of anesthesia, the CPOM monitor will be secured to the temporal region of the participant's forehead to measure and record the cerebral hemodynamic data before, during, and following intubation. Hemodynamic, respiratory, body temperature, and anesthetic data will be continuously digitally records. The CPOM device will be detached after extubation in the operative room.

SUMMARY:
This study uses a CPOM Optical neuromonitor to assess the relationship between brain cytochrome C oxidase, cerebral oxygen saturation and blood pressure during surgery performed under general anesthesia.

DETAILED DESCRIPTION:
During various surgical procedures, blood supply to the brain can be jeopardized either due to interruption of flow as occurs during carotid surgery, or due to inadequate arterial pressure which can occur in settings as diverse as heart surgery or shoulder surgery. This is a prospective observational study of brain oxygen levels, brain metabolism and blood pressure in 50 adult surgical patients under general anesthesia using a CPOM Optical neuromonitor.

This is an observational study. The primary objective of this study is to describe the changes in redox state of brain CCO (reflecting oxidative metabolism), CBFi, and brain tissue oxygen saturation in relation to systemic blood pressure in patients during general anesthesia/cardiopulmonary bypass (CPB). This study represents the first opportunity to assess this combined technology in adult patients and will provide important data to support further investigations in brain-at-risk patients.

These 50 patients will be used to help the investigators to obtain pilot data about the relationship between brain cytochrome C oxidase (bCCO), cerebral oxygen saturation (ScO2), and blood pressure (especially hypotension) using a CPOM device. Cerebral auto regulation indices will also be determined. No intervention will be applied.

ELIGIBILITY:
Inclusion Criteria:

* All adult surgical patients (>18 year-old) who require general anesthesia for their surgery
* Patients required an arterial line for his/her procedure

Exclusion Criteria:

* Emergency surgery
* Unable to obtain consent
* Condition that preclude the use of CPOM monitor (e.g. skin lesion in the forehead)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted for surgery requiring general anesthesia and required to have an arterial line.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Brain cytochrome C oxidase level. | Intraoperative
  The cytochrome C oxidase level which reflects the brain oxidative metabolism will be measured by a CPOM Optical Neuromonitor.
Brain saturation (ScO2) | Intraoperative
  The brain saturation (ScO2) (%) will be measured by a CPOM Optical Neuromonitor.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chui, MBChB, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Bale G, Elwell CE, Tachtsidis I. Errata: From Jobsis to the present day: a review of clinical near-infrared spectroscopy measurements of cerebral cytochrome-c-oxidase. J Biomed Opt. 2016 Sep;21(9):099801. doi: 10.1117/1.JBO.21.9.099801. No abstract available. PMID 27411110
- [Background] de Roever I, Bale G, Cooper RJ, Tachtsidis I. Functional NIRS Measurement of Cytochrome-C-Oxidase Demonstrates a More Brain-Specific Marker of Frontal Lobe Activation Compared to the Haemoglobins. Adv Exp Med Biol. 2017;977:141-147. doi: 10.1007/978-3-319-55231-6_19. PMID 28685438
- [Background] Rajaram A, Bale G, Kewin M, Morrison LB, Tachtsidis I, St Lawrence K, Diop M. Simultaneous monitoring of cerebral perfusion and cytochrome c oxidase by combining broadband near-infrared spectroscopy and diffuse correlation spectroscopy. Biomed Opt Express. 2018 May 10;9(6):2588-2603. doi: 10.1364/BOE.9.002588. eCollection 2018 Jun 1. PMID 30258675
- [Background] Diop M, Kishimoto J, Toronov V, Lee DS, St Lawrence K. Development of a combined broadband near-infrared and diffusion correlation system for monitoring cerebral blood flow and oxidative metabolism in preterm infants. Biomed Opt Express. 2015 Sep 10;6(10):3907-18. doi: 10.1364/BOE.6.003907. eCollection 2015 Oct 1. PMID 26504641
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Davie SN, Grocott HP. Impact of extracranial contamination on regional cerebral oxygen saturation: a comparison of three cerebral oximetry technologies. Anesthesiology. 2012 Apr;116(4):834-40. doi: 10.1097/ALN.0b013e31824c00d7. PMID 22343469
- [Background] Ogoh S, Sato K, Okazaki K, Miyamoto T, Secher F, Sorensen H, Rasmussen P, Secher NH. A decrease in spatially resolved near-infrared spectroscopy-determined frontal lobe tissue oxygenation by phenylephrine reflects reduced skin blood flow. Anesth Analg. 2014 Apr;118(4):823-9. doi: 10.1213/ANE.0000000000000145. PMID 24651237
- [Background] Murkin JM. Is it better to shine a light, or rather to curse the darkness? Cerebral near-infrared spectroscopy and cardiac surgery. Eur J Cardiothorac Surg. 2013 Jun;43(6):1081-3. doi: 10.1093/ejcts/ezt186. Epub 2013 Mar 29. No abstract available. PMID 23543201
- [Background] Olesen ND, Sorensen H, Ambrus R, Svendsen LB, Lund A, Secher NH. A mesenteric traction syndrome affects near-infrared spectroscopy evaluated cerebral oxygenation because skin blood flow increases. J Clin Monit Comput. 2018 Apr;32(2):261-268. doi: 10.1007/s10877-017-0014-2. Epub 2017 Mar 14. PMID 28293809
- [Background] Bainbridge A, Tachtsidis I, Faulkner SD, Price D, Zhu T, Baer E, Broad KD, Thomas DL, Cady EB, Robertson NJ, Golay X. Brain mitochondrial oxidative metabolism during and after cerebral hypoxia-ischemia studied by simultaneous phosphorus magnetic-resonance and broadband near-infrared spectroscopy. Neuroimage. 2014 Nov 15;102 Pt 1:173-83. doi: 10.1016/j.neuroimage.2013.08.016. Epub 2013 Aug 17. PMID 23959202
- [Background] Tisdall MM, Tachtsidis I, Leung TS, Elwell CE, Smith M. Increase in cerebral aerobic metabolism by normobaric hyperoxia after traumatic brain injury. J Neurosurg. 2008 Sep;109(3):424-32. doi: 10.3171/JNS/2008/109/9/0424. PMID 18759572
- [Background] Diop M, Verdecchia K, Lee TY, St Lawrence K. Calibration of diffuse correlation spectroscopy with a time-resolved near-infrared technique to yield absolute cerebral blood flow measurements. Biomed Opt Express. 2011 Jul 1;2(7):2068-81. doi: 10.1364/BOE.2.002068. Epub 2011 Jun 28. PMID 21750781
- [Background] Durduran T, Yodh AG. Diffuse correlation spectroscopy for non-invasive, micro-vascular cerebral blood flow measurement. Neuroimage. 2014 Jan 15;85 Pt 1(0 1):51-63. doi: 10.1016/j.neuroimage.2013.06.017. Epub 2013 Jun 14. PMID 23770408
- [Background] Murkin JM, Kamar M, Silman Z, Balberg M, Adams SJ. Intraoperative Cerebral Autoregulation Assessment Using Ultrasound-Tagged Near-Infrared-Based Cerebral Blood Flow in Comparison to Transcranial Doppler Cerebral Flow Velocity: A Pilot Study. J Cardiothorac Vasc Anesth. 2015 Oct;29(5):1187-93. doi: 10.1053/j.jvca.2015.05.201. Epub 2015 May 27. PMID 26384626
- [Background] McManus R, Froats E, St Lawrence K, Vanuum S, Diop M. Dynamic Relationship between Cerebral Blood Flow and Symptoms of Hypoglycemia. Canadian Journal of Diabetes 42(5): S12, 2018.
- [Background] Govier AV, Reves JG, McKay RD, Karp RB, Zorn GL, Morawetz RB, Smith LR, Adams M, Freeman AM. Factors and their influence on regional cerebral blood flow during nonpulsatile cardiopulmonary bypass. Ann Thorac Surg. 1984 Dec;38(6):592-600. doi: 10.1016/s0003-4975(10)62316-8. PMID 6439135
- [Background] Lundar T, Froysaker T, Lindegaard KF, Wiberg J, Lindberg H, Rostad H, Nornes H. Some observations on cerebral perfusion during cardiopulmonary bypass. Ann Thorac Surg. 1985 Apr;39(4):318-23. doi: 10.1016/s0003-4975(10)62621-5. PMID 3985707
- [Background] Verdecchia K, Diop M, Lee A, Morrison LB, Lee TY, St Lawrence K. Assessment of a multi-layered diffuse correlation spectroscopy method for monitoring cerebral blood flow in adults. Biomed Opt Express. 2016 Aug 24;7(9):3659-3674. doi: 10.1364/BOE.7.003659. eCollection 2016 Sep 1. PMID 27699127